CLINICAL TRIAL: NCT01568684
Title: Pharmacogenetics and Neuroimaging in Major Depressive Disorder (PAN-D)
Brief Title: Brain Imaging, Genetics and Treatment for Major Depression
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120099; 12-M-0099
Record Dates: First submitted 2012-03-30; First posted 2012-04-02 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2012-12-11

CONDITIONS: Depressive Disorder; Depressive Disorder, Major; Depression
Keywords: Magnetic Resonance Spectroscopy; Depression; Depression Treatment; Major Depression; Unipolar Depression
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Depression | interventions — Citalopram

INTERVENTIONS:
Other: Citalopram — Treatment

SUMMARY:
Background:

- Antidepressants help many people with depression, however, some do not seem to benefit as much. Currently, it is not possible to determine who will improve with certain antidepressants. Studies have shown that genes may influence whether an antidepressant works for an individual. Other studies have shown that depressed people tend to have lower levels of a chemical called glutamate in parts of their brain, and that glutamate levels increase after recovering from depression. Researchers want to study the antidepressant citalopram (Celexa) to see how it affects glutamate levels in the brain. They also want to study how a person s genes affect their response to this treatment.

Objectives:

- To see whether glutamate levels and certain genes affect how a person responds to a particular antidepressant medication.

Eligibility:

- Individuals between 25 and 55 years of age who have been diagnosed with major depression (without psychotic features). Participants may not have tried more than three antidepressant treatments.

Design:

* Participants will be screened with a physical exam and medical history. They will answer questions about mood and current feelings of depression, as well as family history of depression. Blood and urine samples will be collected.
* This study will have two phases. The first phase may last up to 7 weeks depending on current antidepressant use and involves one to seven outpatient visits. The second phase lasts 8 weeks and involves five outpatient visits, one every 2 weeks.
* In the first phase, participants will stop taking their current antidepressant medications for at least 2 weeks before the next phase of the study. Participants who are on fluoxetine (Prozac) will need to be off it for 6 weeks.
* At the end of this phase, participants will have brain imaging studies to look at brain function and chemistry.
* In the second phase, participants will take citalopram at the standard dose. They will answer questions about mood and response to the medication. They will also provide blood and saliva samples for tests.
* At the end of this phase, participants will have brain imaging studies to look at brain function and chemistry.

DETAILED DESCRIPTION:
Objective:

Major depressive disorder (MDD) is a serious, debilitating, life-shortening illness that affects many persons of all ages and backgrounds. Although many patients suffering from MDD can expect improvement with antidepressant treatment, only a minority experience full remission, and little is known about the basis for individual differences in treatment outcome. The rationale for this study follows from the findings that treatment response in major depression is associated with: 1) variation in the genes encoding the serotonin 2A receptor (HTR2A) and the KA1 subunit of the glutamate-kainate receptor (GRIK4); and 2) increases in prefrontal glutamate/glutamine (glx) concentration measured by [+H] magnetic resonance spectroscopy (MRS). The central hypothesis is that genes associated with citalopram treatment outcome modulate glutamate concentrations in prefrontal brain (PFB) and thus facilitate response to citalopram treatment. Such information is important because it would ultimately allow the development of better treatments for MDD.

Study population:

A total of 104 moderate to severe MDD outpatients aged 25-55 with a baseline 17-item Hamilton Depression Rating Scale (HDRS) score of greater than or equal to18 who meet DSM-IV criteria for non-psychotic major depressive disorder (MDD) will be enrolled in the course of the study.

Design:

Subjects will be screened with an on-site research psychiatric evaluation using a structured interview (MINI plus). After screening, participants will provide a DNA sample, which will be analyzed to determine the patient s genotype at several relevant loci. All patients will then complete an eight-week period of citalopram treatment, during which time they will be evaluated bi-weekly with self-report questionnaires and clinician ratings to determine change of MDD symptoms. Participants will also undergo pre- and post-treatment MRS scans to determine glutamate concentration in the prefrontal brain.

Treatment outcome measures:

The Quick Inventory of Depressive Symptomatology - Clinician-Rated (QIDS-C16) will be the primary clinical outcome measure and will be collected at baseline and at each treatment visit. Additionally, levels of glutamate in the prefrontal regions of the brain will be measured by MRS. Clinical response will be defined as a decrease of 50 percent or greater in QIDS-C16 score from baseline, and remission will be defined as a QIDS-C16 score of less than 6.

This proposal is part of a K99 training grant and has undergone extensive external review (K99MH085098-01A2).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male and female subjects aged between 25 and 55 years
* Score of 18 or higher on the 17-item Hamilton Depression Rating Scale (HDRS17). We have set the HDRS17 cutoff score to greater than or equal to18 to increase the contrast signals between remitters and non-remitters, MRS imaging and genotypic groups.
* Meets DSM-IV criteria for chronic or recurrent non-psychotic MDD
* No more than 3 failed FDA-approved antidepressant treatments within the current episode
* No alcohol use in the last 7 days
* Fluent in English or Spanish
* Capacity to understand the nature of the study and provide informed consent

EXCLUSION CRITERIA:

* Lifetime history of schizophrenia, schizoaffective disorder or psychosis not otherwise specified
* Lifetime history of bipolar disorder (I, II, or not otherwise specified)
* Lifetime history of anorexia nervosa or bulimia nervosa
* Current primary obsessive-compulsive disorder (OCD)
* History of intolerability to citalopram
* Lack of response to an adequate trial of citalopram or escitalopram in the current or previous episodes of MDD
* Have failed to respond to more than three antidepressants during current major depressive episode
* Lack of response to 7 or more sessions of ECT in the current or previous episodes of MDD
* Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease
* Females who are sexually active and who are not willing to use effective contraception for 8-weeks while participating in this study or are pregnant or breast feeding
* Concomitant medication use which contraindicates the use of the study medication
* Requires any of the following exclusionary medications: antipsychotic medications, anticonvulsant medications, antidepressant medications, mood stabilizers, central nervous system stimulants
* Patients on thyroid medication for hypothyroidism: stable on thyroid medication for < 2 months
* Current participation in any modality of psychotherapy and the patient is not willing to forgo it during participation
* Have a history of drug or alcohol dependence or current abuse within the last 3 months
* Past history of significant head injury with loss of consciousness for about 24 hours or more
* Current or past history of seizure disorder
* Suicidal ideation with plan and/or intent
* Have received any investigational drug within the last 30 days
* Metallic (ferromagnetic) implants, including pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pump, shrapnel fragments, and possible small metal fragments in the eye
* Unable to lie flat on back for up to 2 hours
* Claustrophobia in scanner
* Positive drug screen
* HIV-positive.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03-12; Primary Completion 2012-12-11 (Actual); Study Completion 2012-12-11 (Actual)

PRIMARY OUTCOMES:
Changes in prefrontal glutamate concentration after citalopram treatment.

SECONDARY OUTCOMES:
Changes in depressive symptoms after citalopram treatment.
Association between glutamate changes and genetic variation.

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Laje, M.D., Principal Investigator — National Institute of Mental Health (NIMH)

REFERENCES:
- [Background] Caetano SC, Fonseca M, Olvera RL, Nicoletti M, Hatch JP, Stanley JA, Hunter K, Lafer B, Pliszka SR, Soares JC. Proton spectroscopy study of the left dorsolateral prefrontal cortex in pediatric depressed patients. Neurosci Lett. 2005 Aug 26;384(3):321-6. doi: 10.1016/j.neulet.2005.04.099. PMID 15936878
- [Background] Cho MK. Understanding incidental findings in the context of genetics and genomics. J Law Med Ethics. 2008 Summer;36(2):280-5, 212. doi: 10.1111/j.1748-720X.2008.00270.x. PMID 18547195
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508